CLINICAL TRIAL: NCT04416841
Title: Efficacy of Tai Chi Chuan on Cognitive Function in Type 2 Diabetes Mellitus Patients Accompanied With Mild Cognitive Impairment
Brief Title: Tai Chi Chuan as Rehabilitation Program for Mild Cognitive Impairment in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jing Tao (Other)
Collaborators: Second Affiliated Hospital of Heilongjiang University of Chinese Medicine (Other); Bao'an District People's Hospital of Shenzhen (Unknown); Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); Peking University (Other); University of Electronic Science and Technology of China (Other)
Responsible Party: Sponsor-Investigator, Jing Tao, PhD, Fujian University of Traditional Chinese Medicine
Organization: Fujian University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FujianUTCM
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus, Type 2; Cognitive Dysfunction
Keywords: Tai Chi Chuan; Cognitive Function; Postural Balance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tai Chi Chuan Group (Experimental): In addition to conventional medical treatment, participants will receive 3 sessions of 1-hour Tai Chi Chuan training per week for 24 weeks and standard diabetic care education.
  Interventions: Behavioral: Tai Chi Chuan
- Fitness Walking Group (Active Comparator): In addition to conventional medical treatment, participants will receive 3 sessions of 1-hour fitness walking training per week for 24 weeks and standard diabetic care education
  Interventions: Behavioral: Fitness Walking
- Control group (Other): In addition to conventional medical treatment, participants will receive standard diabetic care education 0.5hour/session, 2 sessions/month for 6 months.
  Interventions: Behavioral: Standard Diabetic Care Education

INTERVENTIONS:
Behavioral: Tai Chi Chuan — Participants would take 24-form simplified Tai Chi Chuan 1 hour/session, 3sessions/week for 24 weeks. There were 10 minutes warm-up, 40 minutes Tai Chi Chuan lesson and 10 minutes cool-down exercises in the Tai Chi Chuan training. Besides, they would also take standard diabetic care education 0.5hour/session, 2 sessions/month for 6 months.
  Arms: Tai Chi Chuan Group
Behavioral: Fitness Walking — Participants would take fitness walking training 1 hour/session, 3sessions/week for 24 weeks. There were 10 minutes warm-up, 40 minutes fitness walking and 10 minutes cool-down exercises in the fitness walking training, the exercise intensity was 50% to 70% of the maximum heart rate. Besides, they would also take standard diabetic care education 0.5hour/session, 2 sessions/month for 6 months.
  Arms: Fitness Walking Group
Behavioral: Standard Diabetic Care Education — Participants would take standard diabetic care education 0.5hour/session, 2 sessions/month for 6 months.
  Arms: Control group

SUMMARY:
The patients with type 2 diabetes mellitus (T2DM) is expected to rise to 439 million in 2030, accounting for 7.7% the population in the world. There are nearly 10 million T2DM patients with mild cognitive impairment (MCI) among people over 65 years old , accounting for about 8% of the people over 65 years old in China. The medical cost for patients with T2DM/MCI is 2.5 to 4 times higher than those without T2DM. And T2DM will increase the risk of cognitive impairment, and lead to various complications which will bring serious social and medical economic burden.

DETAILED DESCRIPTION:
It is critically important to identify effective treatments to enhance functional status of T2DM/MCI patients. Exercise has been shown to be beneficial for T2DM/MCI patients. As a Chinese traditional mind-body exercise that consists of both physical and mediation components, Tai Chi Chuan has been proved to be helpful in global cognition, memory, executive function and attention of MCI, and blood sugar of T2DM. However, the evidence of the effect of Tai Chi Chuan on T2DM/MCI patients is limited. The purpose of this study is to explore the effect of Tai Chi Chuan treating T2DM/MCI patients in cognitive function, balance, motor and sensation function, blood sugar, biochemistry profile and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. clinician diagnosis of T2DM;
2. presence of mild cognitive impairment, not demented;
3. age ≥ 60 years old;
4. did not engage in regular exercise in the last three months (at least 3 times a week, at least 20 minutes of regular exercise each time);
5. informed consent and voluntary participation.

Exclusion Criteria:

1. cognitive impairment caused by other reasons, taking drugs, poisoning, etc;
2. presence of medical conditions that unable or unsafe to exercise, such as depression symptoms, uncontrolled hypertension/ blood pressure/ blood glucose, nervous system diseases(stroke, Parkinson's disease, etc), musculoskeletal system diseases(arthritis, history of hip and/or knee joint replacement, etc), etc;
3. participating in other experiments that influence this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Global cognition-Montreal Cognitive Assessment at 36 Weeks | 36 weeks (post-intervention follow-up)
  Montreal Cognitive Assessment

SECONDARY OUTCOMES:
Global cognition-Montreal Cognitive Assessment at 24 weeks | 24 weeks (post-intervention)
  Montreal Cognitive Assessment
Memory function-Wechsler Memory Scale at 24, 36 Weeks | 24, 36 weeks
  Wechsler Memory Scale
Digital Symbol test at 24, 36 weeks | 24, 36 weeks
  Digital Symbol test
Trial Making Test part B at 24, 36 weeks | 24, 36 weeks
  Trial Making Test part B
Stroop color word test at 24, 36 weeks | 24, 36 weeks
  Stroop color word test
Boston naming test at 24, 36 weeks | 24, 36 weeks
  Boston naming test
Rey-Osterrieth complex graphics test at 24, 36 weeks | 24, 36 weeks
  Rey-Osterrieth complex graphics test
Multi-task balance test: Time up and go test; Time up and go test + cognitive task;Time up and go test + motor task;Time up and go test + cognitive task + motor task at 24, 36 weeks | 24, 36 weeks
  Time up and go test; Time up and go test + cognitive task (animal naming); Time up and go test + motor task (holding a cup of water); Time up and go test + cognitive task + motor task.
Functional reach test at 24, 36 weeks | 24, 36 weeks
  Functional reach test
One leg stance test at 24, 36 weeks | 24, 36 weeks
  One leg stance test
Grip strength at 24, 36 weeks | 24, 36 weeks
  Grip strength
Five times sit-to-stand test at 24, 36 weeks | 24, 36 weeks
  Five times sit-to-stand test
Sensation function at 24, 36 weeks | 24, 36 weeks
  Tactile sensation; Two-point discrimination sensation; Vibration sensation.
Fall efficiency-Modified Falls Efficacy Scale at 24, 36 weeks | 24, 36 weeks
  Modified Falls Efficacy Scale
Quality of life-Medical Outcomes Study 36-item Short-Form Health Survey at 24, 36 weeks | 24, 36 weeks
  Medical Outcomes Study 36-item Short-Form Health Survey (SF-36)

OTHER OUTCOMES:
Blood glucose metabolism index at 24, 36 weeks | 24, 36 weeks
  fasting blood glucose; glycosylated hemoglobin; fasting insulin
Blood lipid metabolism index at 24, 36 weeks | 24, 36 weeks
  total cholesterol (TC); total triglyceride (TG); low density lipoprotein (LDL),;high density lipoprotein (HDL).
Circulating levels of AGE and sRAGE at 24, 36 weeks | 24, 36 weeks
  Circulating levels of AGE and sRAGE
functional Magnetic Resonance Imaging (fMRI) | baseline, 24 weeks
  functional Magnetic Resonance Imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian University of Traditional Chinese Medicine, Fuzhou, Fujian, China

REFERENCES:
- [Background] You Y, Liu Z, Chen Y, Xu Y, Qin J, Guo S, Huang J, Tao J. The prevalence of mild cognitive impairment in type 2 diabetes mellitus patients: a systematic review and meta-analysis. Acta Diabetol. 2021 Jun;58(6):671-685. doi: 10.1007/s00592-020-01648-9. Epub 2021 Jan 8. PMID 33417039
- [Background] Qin J, Chen Y, Guo S, You Y, Xu Y, Wu J, Liu Z, Huang J, Chen L, Tao J. Effect of Tai Chi on Quality of Life, Body Mass Index, and Waist-Hip Ratio in Patients With Type 2 Diabetes Mellitus: A Systematic Review and Meta-Analysis. Front Endocrinol (Lausanne). 2021 Jan 19;11:543627. doi: 10.3389/fendo.2020.543627. eCollection 2020. PMID 33542702
- [Background] Guo S, Xu Y, Qin J, Chen Y, You Y, Tao J, Liu Z, Huang J. Effect of tai chi on glycaemic control, lipid metabolism and body composition in adults with type 2 diabetes: A meta-analysis and systematic review. J Rehabil Med. 2021 Mar 22;53(3):jrm00165. doi: 10.2340/16501977-2799. PMID 33594445
- [Background] Bai A, Tao L, Huang J, Tao J, Liu J. Effects of physical activity on cognitive function among patients with diabetes in China: a nationally longitudinal study. BMC Public Health. 2021 Mar 11;21(1):481. doi: 10.1186/s12889-021-10537-x. PMID 33706749
- [Background] Yin L, Qin J, Chen Y, Xie J, Hong C, Huang J, Xu Y, Liu Z, Tao J. Impact of Body Mass Index on Static Postural Control in Adults With and Without Diabetes: A Cross-Sectional Study. Front Endocrinol (Lausanne). 2021 Dec 24;12:768185. doi: 10.3389/fendo.2021.768185. eCollection 2021. PMID 35002958
- [Background] Xie J, Yin L, Huang J, Xu Y, Chen Y, Qin J, Liu Z, Tao J. Correlation between impaired hemodynamic response and cardiopulmonary fitness in middle-aged type 2 diabetes mellitus patients: a case-control study. Eur J Appl Physiol. 2022 Oct;122(10):2295-2303. doi: 10.1007/s00421-022-05008-z. Epub 2022 Jul 20. PMID 35859047
- [Derived] Chen Y, Qin J, Tao L, Liu Z, Huang J, Liu W, Xu Y, Tang Q, Liu Y, Chen Z, Chen S, Liang S, Chen C, Xie J, Liu J, Chen L, Tao J. Effects of Tai Chi Chuan on Cognitive Function in Adults 60 Years or Older With Type 2 Diabetes and Mild Cognitive Impairment in China: A Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e237004. doi: 10.1001/jamanetworkopen.2023.7004. PMID 37022680